CLINICAL TRIAL: NCT00954798
Title: Immunogenicity and Safety of Multiple Formulations of an Intramuscular Inactivated, Split Virion Swine-origin A/H1N1 Influenza Vaccine With and Without Adjuvant in Healthy European Adult and Elderly Subjects
Brief Title: A Study of Swine-origin A/H1N1 Influenza Vaccines in Healthy European Adults and the Elderly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GPF07; UTN: U1111-1111-4918; 2009-013344-37 (EudraCT Number)
Record Dates: First submitted 2009-08-03; First posted 2009-08-07 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Influenza; Swine-origin A/H1N1 Influenza
Keywords: Influenza; Pandemic Flu; Swine-origin Influenza; Inactivated split-virion vaccine; Adjuvant; Adult
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A/H1N1 Vaccine Group 1 (Experimental): All participants will receive A/H1N1 vaccine formulation 1 at Visits 1 and 2; a subset will receive a trivalent influenza vaccine (TIV) at Month 13.
  Interventions: Biological: Swine A/H1N1 influenza vaccine (split virion, inactivated)
- A/H1N1 Vaccine Group 2 (Experimental): All participants will receive A/H1N1 vaccine formulation 2 at Visits 1 and 2; a subset will receive a trivalent influenza vaccine (TIV) at Month 13.
  Interventions: Biological: Swine A/H1N1 influenza vaccine (split virion, inactivated)
- A/H1N1 Vaccine Group 3 (Experimental): Participants will receive A/H1N1 vaccine formulation 3
  Interventions: Biological: Swine A/H1N1 influenza vaccine (split virion, inactivated)

INTERVENTIONS:
Biological: Swine A/H1N1 influenza vaccine (split virion, inactivated) — 0.5 mL, Intramuscular on Day 0 and day 21 (all participants); and 0.5 mL of trivalent influenza vaccine (TIV) at Month 13 (antibody persistence subset)
  Arms: A/H1N1 Vaccine Group 1
Biological: Swine A/H1N1 influenza vaccine (split virion, inactivated) — 0.5 mL, Intramuscular on Day 0 and day 21 (all participants), and 0.5 mL of trivalent influenza vaccine (TIV) at Month 13 (antibody persistence subset).
  Arms: A/H1N1 Vaccine Group 2
Biological: Swine A/H1N1 influenza vaccine (split virion, inactivated) — 0.5 mL, Intramuscular on Day 0 and Day 21
  Arms: A/H1N1 Vaccine Group 3

SUMMARY:
The purpose of this study is to generate data on immunogenicity and safety of the monovalent H1N1 vaccine in support of the development and registration.

Primary objectives:

* To describe the immune response to study vaccine 21 days after each vaccination.
* To describe the antibody persistence 8 months after the first vaccine administration using hemagglutination inhibition (HAI) method in a randomized subset of adult subjects who received two injections.
* To describe the immune response against the A/H1N1 strain using HAI method 21 days after a vaccination with the 2010-2011 Northern Hemisphere (NH) seasonal trivalent influenza vaccine (TIV) administered 13 months after the first vaccination in a subset subjects who received the A/H1N1 influenza vaccine and in subjects naïve to the swine origin A/H1N1 strain.
* To describe the safety profiles of study vaccines in all participants.

DETAILED DESCRIPTION:
All participants will receive two injections of their randomized vaccine on Day 0 and Day 21, respectively.

A subset of the participants will receive a third vaccine injection (2010-2011 Northern Hemisphere [NH] seasonal trivalent influenza vaccine [TIV]) approximately 13 months after the first vaccination; additionally, a subset of participants' naïve to the swine-origin A/H1N1 strain will also receive one vaccine injection of the 2010-2011 NH seasonal TIV.

ELIGIBILITY:
Inclusion Criteria :

* Aged 18 years or over on the day of inclusion
* Informed Consent Form has been signed and dated
* Able to attend all scheduled visits and to comply with all trial procedures
* For a woman of childbearing potential, use of an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination until at least 4 weeks after the last vaccination
* Entitled to national social security

At Visit 05, for antibody persistence assessment:

* Addendum 1 to Informed Consent Form has been signed and dated
* Having received two vaccinations with the vaccine formulation 1 or 2.

At Month 13, for trivalent influenza vaccine (TIV) administration in subjects who received the A/H1N1 influenza vaccine:

- Addendum 2 to Informed Consent Form has been signed and dated

Exclusion Criteria :

* Known pregnancy, or a positive urine pregnancy test
* Currently breastfeeding a child
* Participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the first trial vaccination
* Planned participation in another clinical trial during the present trial period
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination
* Planned receipt of any vaccine prior to the Day 42 blood sample
* Receipt of blood or blood-derived products in the past 3 months, which might interfere with assessment of the immune response
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Self-reported seropositivity for Human Immunodeficiency Virus (HIV), Hepatitis B, or Hepatitis C
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine(s) used in the trial or to a vaccine containing any of the same substances
* Self-reported thrombocytopenia, contraindicating intramuscular (IM) vaccination
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction that might interfere with the ability to comply with trial procedures
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion
* Employee of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as family members of the employees or the Investigator
* Previous participation in a trial investigating a vaccine with the swine-origin A/H1N1 influenza strain
* Confirmed infection with the swine-origin A/H1N1 influenza strain (different from the seasonal strain) in 2009
* Febrile illness (temperature ≥ 38.0°C) or moderate or severe acute illness/infection on the day of vaccination, according to Investigator judgment
* Receipt of any allergy shots and/or seasonal allergy medication in the 7-day period prior to enrollment (vaccination), or scheduled to receive any allergy shots and/or seasonal allergy medication in the 7-day period after enrollment (vaccination)

At Month 8, for antibody persistence assessment:

- Subjects who received, in the context of a pandemic immunization program, another A/H1N1 pandemic influenza vaccine than the Investigational Medicinal Products.

Additional criteria for subset to receive only the TIV:

* History of pandemic A/H1N1 influenza vaccination
* History of clinically or laboratory confirmed pandemic A/H1N1 influenza infection
* Receipt of an adjuvanted influenza vaccine in a clinical trial within the previous 12 months
* Planned receipt of any vaccine during the present trial period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2009-08; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the immunogenicity of Swine A/H1N1 influenza vaccine | 21 days post-vaccination
To provide information concerning the safety in terms of solicited injection site and systemic reactions following vaccination with Swine A/H1N1 influenza vaccine | 0 to7 days post-vaccination and entire study duration

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (6):
- France (6):
  - Angers
  - Château-Gontier
  - Cherbourg
  - Équeurdreville-Hainneville
  - Laval
  - Tiercé

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com